CLINICAL TRIAL: NCT01755338
Title: Effect of Steroids on Cerebrospinal Fluid Markers of Inflammation and Neuronal Damage After Surgical Aortic Valve Replacement
Brief Title: Effect of Steroids on Cerebral Inflammation and Neuronal Damage After Surgical Aortic Valve Replacement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Mattias Danielson, MD, Sahlgrenska University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2012-004232-37
Record Dates: First submitted 2012-12-18; First posted 2012-12-24 (Estimated); Last update posted 2017-06-01 (Actual); Status verified 2017-05

CONDITIONS: Aortic Stenosis
Keywords: cerebrospinal fluid; inflammatory markers; heart surgery; neuronal damage; blood brain barrier
MeSH Terms: conditions — Aortic Valve Stenosis | interventions — Methylprednisolone; Methylprednisolone Hemisuccinate; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Methylprednisolone (Active Comparator): Methylprednisolone i.v. 15mg/kg x 1 intraoperative Aortic Valve Replacement
  Interventions: Drug: Methylprednisolone
- Placebo (NaCl) (Placebo Comparator): Placebo i.v., x1, intraoperative Aortic Valve Replacement
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Methylprednisolone — Methylprednisolone 15mg/kg
  Other Names: Solu-Medrol
  Arms: Methylprednisolone
Drug: Placebo — Placebo
  Other Names: Sodium Chloride
  Arms: Placebo (NaCl)

SUMMARY:
The purpose of this study is to investigate if methylprednisolone is effective in reducing the cerebral inflammatory response after open heart surgery with cardiopulmonary bypass.

DETAILED DESCRIPTION:
In a previous study we found that patients undergoing aortic valve surgery had elevated cerebrospinal inflammatory markers. In this study we aim to investigate if this inflammatory response can be reduced after treatment with steroids.

30 patients will be randomized to intraoperative treatment with either placebo or methylprednisolone 15mg/kg. CSF and blood will be collected the day before and the day after surgery, analyzed for markers of inflammation (IL-6, IL-8), neuronal damage (S-100) and blood brain barrier function (alb).

ELIGIBILITY:
Inclusion Criteria:

* elective aortic surgery +/- coronary artery bypass grafting (CABG)

Exclusion Criteria:

* coagulopathy
* preoperative neurologic deficit
* uncontrolled hypertension

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-12; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Changes in cerebrospinal fluid (CSF) levels of IL-6, IL-8, S100B, alb | 24h after surgery

SECONDARY OUTCOMES:
Postoperative/intraoperative insulin demand | 24h after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Sven-Erik Ricksten, Professor, Study Chair — Sahlgrenska University Hospital
Locations (1):
- Sahlgrenska University Hospital, Gothenburg, VGR, Sweden

REFERENCES:
- [Derived] Danielson M, Reinsfelt B, Westerlind A, Zetterberg H, Blennow K, Ricksten SE. Effects of methylprednisolone on blood-brain barrier and cerebral inflammation in cardiac surgery-a randomized trial. J Neuroinflammation. 2018 Sep 27;15(1):283. doi: 10.1186/s12974-018-1318-y. PMID 30261896